CLINICAL TRIAL: NCT03429023
Title: Multicenter Observational Study on Epidemiology, Treatment and Outcome of Mucormycosis in India
Brief Title: Descriptive Epidemiology on Management of Mucormycosis
Status: Completed | Type: Observational
Sponsor: Fungal Infection Study Forum (Other)
Collaborators: Mylan India Limited (Unknown)
Responsible Party: Principal Investigator, Arunaloke Chakrabarti, Chairman FISF, Fungal Infection Study Forum
Other Study IDs: FISF 001.3
Record Dates: First submitted 2017-07-29; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Mycoses
Keywords: Mucormycosis
MeSH Terms: conditions — Mycoses; Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational chart review of all patients with confirmed and probable diagnosis of mucormycosis at 19 centers across Indian hospital. Data will collect using a standardized CRF. All collected data will be entered into a database prior to analysis. Broadly data will be collected on demography, clinical characteristics, diagnosis, treatment and outcome for each patient. Patient will continue to receive treatment as per treating physicians advise. Primary outcome for this study will be overall survival at 45 & 90 days.

DETAILED DESCRIPTION:
Introduction

Mucormycosis is a life threatening angio-invasive fungal infection generally occurring in immunocompromised individuals. In recent years the incidence has increased globally and alarmingly in India especially in patients with uncontrolled diabetes. Mucormycosis is associated with very high morbidity and mortality. Mortality can be reduced with increased awareness of the disease, and aggressive medical and surgical intervention. Though few case series of mucormycosis are published from India, multiple gaps in knowledge exist regarding epidemiology, diagnosis and management of the disease in this country. It is therefore proposed to conduct this multicentric observational study in India to evaluate epidemiology, mode of diagnosis, management practices and outcome in patients with mucormycosis.

Study Objectives

Primary:

- To describe the epidemiology, diagnosis, treatment practices and outcome of mucormycosis in India

Secondary:

* Sites involved in mucormycosis
* Underlying disease and risk factors for mucormycosis
* Spectrum of agents causing mucormycosis Ð mode of diagnosis of mucormycosis

Methods: Observation chart review Study Sites: We have assembled a network of health center across India called Mucormycosis Study Network (MSN), which consists of 19 centers across the country. Listed in Appendix 1.

Study design: We propose to conduct a single arm prospective observational study.

Study procedures:

Working definition of Proven & Probable mucormycosis used for this study. Proven case: Presence of fungus in the tissue detected by direct microscopy (KOH, Calcoflor white) and Histopathological examination or from any aspiration /tissue from sterile site.

Probable case: Clinical features of infection in organ-site with presence of mucorale in tissue from non-sterile infected site.

Post enrollment, all patients will receive treatment as per the discretion of treating physicians or local hospital protocol. Data on patients' clinical features, risk factors, laboratory and radiological findings will be collected on standardize case report forms (CRF).

Specifically, the extent of disease will be evaluated with appropriate radiological evaluation CT scan/ MRI (Brain, PNS, Thorax, abdomen etc.) Attempt will be made to collect follow up data till 6 months after diagnosis unless the patient lost in follow up or died before six months. All culture isolates will be sent to Mycology Reference Laboratory at PGIMER, Chandigarh for final identification and drug susceptibility testing. Blocks of histopathological specimen will be sent at reference mycology laboratory for patients with histopathological diagnosis of mucormycosis for DNA extraction and species identification.

Primary outcome

1. Overall survival at 45 & 90 days
2. Cure: defined as complete resolution of clinical, radiological and mycological evidence
3. Improved: Resolution of clinical features, radiological regression

Secondary outcomes

1. Grade III and IV toxicities of antifungal agents (Refer Appendix 2 for definition)

Data Collection Data will collect using a standardized CRF. All collected data will be entered into a database prior to analysis. Broadly data will be collected on demography, clinical characteristics, diagnosis, treatment and outcome for each patient.

Patient characteristics: Demographics, Comorbidities (Diabetes, Solid organ Transplant, GVHD requiring steroids, Febrile neutropenia, prolong neutropenia + Steroid therapy, Voriconazole exposure, Immunocompetent patient, Nosocomial [Surgical site, wooden spatula, ECG lead etc], history of road traffic accidents, tsunami, hurricane, Patients receiving immunosuppressives for collagen diseases, Use of monoclonal antibodies for treatment of variety of medical conditions, Iron overload and desferioxamine therapy, Burns patients), Organ dysfunction, Bacterial super infections

Disease characteristics: Site of disease (pulmonary, PNS, Brain, skin and soft tissue, GI, Renal etc), number of lesions, species of mucormycosis

Treatment:

1. . Time to start antifungal drug after (a). Onset of disease i.e. first symptom (b). Diagnosis of mucormycosis
2. . Dose and duration of antifungal agent
3. . Time to Surgical Treatment after (a). Onset of disease i.e. first symptom (b). Diagnosis
4. . Type of Surgical treatment: Radical surgery, Debridement, Repeated debridement Adjuvant treatment used e.g. Deferasirox, posaconazole
5. . Posaconazole maintenance after completion of ABDC

Outcomes:

Overall survival (OS): OS will be measured 2 ways: from onset of first symptoms as reported by patient and from day of admission to last follow-up.

Mortality Related to mucormycosis, not related to Mucormycosis

Treatment Regimen:

The study will not interfere with management at any stage. Treating physician will determine all process of patient management including diagnosis and treatment. Information on antifungal agent used, dosage used and duration of treatment will be collected.

Information on surgical treatment will be collected i.e. time to surgical treatment after diagnosis, debridement, numbers and frequency of debridement, extensive surgical resection.

Control of diabetes, reversal of metabolic parameters, management of immunosuppression will be noted.

Follow up data will also be collected similarly.

Patients will be assessed during hospitalization for drug compliance and toxicities.

Adverse Event will be noted and graded according to standard grading system. Prior and Concomitant Therapy The details of any prior, concomitant or follow up therapy like deferasirox or Posaconazole will also be noted

Statistical Plan Patient, disease and treatment characteristics will be summarized using descriptive statistics. Differences in the primary outcome of survival according to patient, disease and treatment characteristics will be assessed using a log-rank test and illustrated using the Kaplan-Meir analysis. Differences in OS will be summarized as hazard ratio along with 95% confidence intervals (CI). Differences in mortality and toxicities according to patient, disease and treatment characteristics will summarized as risk ratio along with 95% CI. All significance testing will be two sided and set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients regardless of age with a confirmed diagnosis mucormycosis through HPE & /or culture will be enrolled in this study. In suspected cases on histopathology, molecular technique of extraction of DNA from tissue and sequencing to identify the pathogen, will be used to confirm the diagnosis
* All probable cases of mucormycosis.

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 13 hospitals are identified across India for this study. All patients diagnose with confirmed and probable mucormycosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality | Three months after the completion of the study
  Number of deaths

CONTACTS AND LOCATIONS:
Locations (13):
- India (13):
  - Sterling Hospital, Ahmedabad, Gujarat
  - St.Johns Medical College, Bangalore, Karnataka
  - PD Hinduja National Hospital and Medical Research centre, Mumbai, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Gangaram Hospital, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - VMMC and Safdarjung Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Sri Ramachandra Medical College & RI, Chennai, Tamil Nadu
  - Christian Medical College, Vellore, Tamil Nadu
  - Nizams Institute Of Medical Sciences, Hyderabad, Telangana
  - PGIMER, Chandigarh
  - JIPMER, Puducherry